CLINICAL TRIAL: NCT05162066
Title: An Open-Label, Safety, Tolerability, and Proof-of-Concept Study of Oral BCX9930 Therapy in Subjects With Complement 3 Glomerulopathy, Immunoglobulin A Nephropathy, or Primary Membranous Nephropathy
Brief Title: Study to Evaluate the Safety, Tolerability of BCX9930 in Participants With Either Complement 3 Glomerulopathy (C3G), Immunoglobulin A Nephropathy (IgAN), or Primary Membranous Nephropathy (PMN)
Acronym: RENEW
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCX9930-211; 2020-005855-19 (EudraCT Number)
Record Dates: First submitted 2021-11-26; First posted 2021-12-17 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Complement 3 Glomerulopathy; Immunoglobulin A Nephropathy; Membranous Nephropathy
Keywords: BCX9930; factor D inhibitor; oral therapy; Complement 3 Glomerulopathy; Immunoglobulin A Nephropathy; Primary Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative; Glomerulonephritis, IGA; Glomerulonephritis, Membranous

STUDY DESIGN:
Intervention Model Description: Three parallel treatment cohorts based on diagnosis of C3G, IgAN, or PMN. All eligible participants will receive open-label BCX9930.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- C3G cohort (Experimental): Approximately 14 eligible participants with C3G will be enrolled.
  Interventions: Drug: BCX9930
- IgAN cohort (Experimental): Approximately 14 eligible participants with IgAN will be enrolled.
  Interventions: Drug: BCX9930
- PMN cohort (Experimental): Approximately 14 eligible participants with PMN will be enrolled.
  Interventions: Drug: BCX9930

INTERVENTIONS:
Drug: BCX9930 — Administered orally at a dose of 200 mg twice daily for the first 2 weeks, then 400 mg twice daily

SUMMARY:
The objective of this study was to determine the safety and therapeutic potential of BCX9930 in participants with C3G, IgAN, or PMN.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 kilograms (kg)
* Primary diagnosis of C3G, IgAN, or PMN confirmed by central pathology review
* An estimated glomerular filtration rate (eGFR) ≥ 50 milliter per minute per 1.73 meter square (mL/min/1.73 m^2) (or ≥ 30 mL/min/1.73 m^2 after Data Monitoring Committee [DMC] recommendation)
* Receiving treatment with a stable, maximum recommended or maximum tolerated dose of an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) for at least 60 days prior to the Day 1 Visit
* Documentation of current vaccinations against Neisseria meningitidis and Streptococcus pneumoniae or willingness to start vaccination series

Exclusion Criteria:

* Known congenital deficiency of C1s, C1r, C1q, C2, or C4
* History of hematopoietic cell transplant or solid organ transplant or anticipated candidate for transplantation
* Myocardial infarction or cerebrovascular accident within 30 days prior to screening, or current and uncontrolled clinically significant cardiovascular or cerebrovascular condition
* History of malignancy within 5 years prior to the screening visit
* Active serious bacterial, viral, or fungal infection or any other serious infection within 14 days of screening
* Treatment with any systemic immunosuppressive or immunomodulatory therapy within 90 days OR anti-CD20 antibody therapies (eg, rituximab) within 180 days prior to the screening visit
* Treatment with renin inhibitors (eg, aliskiren) or sodium-glucose-cotransporter 2 (SGLT2) inhibitors within 60 days prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla M Nester, MD, MSA, FASN, Principal Investigator — University of Iowa Stead Family Children's Hospital
Locations (11):
- France (2):
  - Investigative Site, Poitiers
  - Investigative Site, Toulouse
- Italy (4):
  - Investigative Site, Bari
  - Investigative Site, Bergamo
  - Investigative Site, Brescia
  - Investigative Site, Turin
- Spain (4):
  - Investigative Site #1, Barcelona
  - Investigative Site #2, Barcelona
  - Investigative Site #1, Madrid
  - Investigative Site #2, Madrid
- Investigative Site, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin J, Radhakrishnan J. What Are Baskets, Umbrellas, and Platforms Doing in Nephrology Clinical Trials? J Am Soc Nephrol. 2025 Feb 3;36(8):1652-1654. doi: 10.1681/ASN.0000000648. No abstract available. PMID 39899371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with either complement 3 glomerulopathy (C3G), immunoglobulin A nephropathy (IgAN), or primary membranous nephropathy (PMN) were planned to be enrolled in the study.
Pre-assignment Details: At the time the study was discontinued, only participants with historical C3G were enrolled.
Groups:
- BCX9930 - C3G Cohort: Participants with complement C3G received BCX9930 tablet orally for up to Day 186 (Week 26).
- BCX9930 - IgAN Cohort: Participants with complement IgAN were to receive BCX9930 tablet orally for up to Day 186 (Week 26).
- BCX9930 - PMN Cohort: Participants with complement PMN were to receive BCX9930 tablet orally for up to Day 186 (Week 26).
Period: Overall Study
Arm/Group | BCX9930 - C3G Cohort | BCX9930 - IgAN Cohort | BCX9930 - PMN Cohort
Started | 2 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Perceived lack of efficacy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BCX9930 - C3G Cohort | BCX9930 - IgAN Cohort | BCX9930 - PMN Cohort | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (16.26) |  |  | 35.5 (16.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  |  | 1
  Male | 1 |  |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 |  |  | 2
  Not Hispanic or Latino | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 2 |  |  | 2
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
24-hour Urine Protein-to-creatinine Ratio (uPCR) [Mean (Standard Deviation); unit: milligram per millimole] — Urinary protein/creatinine ratio (milligram per millimole [mg/mmol]) =urine protein concentration (mg/deciliter [dL])/ urine creatinine concentration (mmol/dL).
  milligram per millimole | 380.5 (137.89) |  |  | 380.5 (137.89)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in 24-hour uPCR at Week 12
Description: Urinary protein/creatinine ratio (mg/mmol) =urine protein concentration (mg/dL)/ urine creatinine concentration (mmol/dL). Decrease of urinary protein/creatinine ratio means improvement of renal disease.
Time Frame: Baseline, Week 12
Population: Safety population with available data was analyzed
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- BCX9930: Participants with complement C3G received BCX9930 tablet orally for up to Day 186 (Week 26).
Arm/Group | BCX9930
Number analyzed (Participants) | 1
percent change | -33.2 (NA) — Standard deviation was not calculated as only one participant was analyzed

2. Primary Outcome: Percent Change From Baseline in 24-hour uPCR at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Safety population with available data was analyzed
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BCX9930
Number analyzed (Participants) | 1
percent change | -8.8 (NA) — Standard deviation was not calculated as only one participant was analyzed

3. Secondary Outcome: Percent Change From Baseline in 24-hour Urinary Protein Excretion
Time Frame: Baseline, Weeks 12, 24,
Population: Safety population with available data was analyzed
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BCX9930
Number analyzed (Participants) | 2
percent change
  Percent Change at Week 12: number analyzed (Participants) | 1
  Percent Change at Week 12 | -40.9 (NA) — Standard deviation was not calculated as only one participant was analyzed
  Percent Change at Week 24: number analyzed (Participants) | 1
  Percent Change at Week 24 | -25.8 (NA) — Standard deviation was not calculated as only one participant was analyzed

4. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate
Description: eGFR was calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula for participants ≥ 18 years old and by the bedside Schwartz formula for participants ≤ 18 years old. eGFR was reported in milliliter per minute per 1.73 per square meter (mL/min/1.73m^2).
Time Frame: Baseline, Weeks 12, 24
Population: Safety population with available data was analyzed
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | BCX9930
Number analyzed (Participants) | 2
mL/min/1.73m^2
  Change at Week 12: number analyzed (Participants) | 1
  Change at Week 12 | -6.0 (NA) — Standard deviation was not calculated as only one participant was analyzed
  Change at Week 24: number analyzed (Participants) | 1
  Change at Week 24 | -5.0 (NA) — Standard deviation was not calculated as only one participant was analyzed

5. Secondary Outcome: Number of Participants With a Treatment-emergent Adverse Event (TEAE)
Description: An Adverse event (AE) was any untoward medical occurrence in a clinical study participant. TEAEs were defined, within a dosing group, as AEs that started on or after the first dose of study treatment through 30 days after the last dose of study drug.
Time Frame: From first dose up to safety follow-up period (Week 28)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930
Number analyzed (Participants) | 2
Participants | 2

6. Secondary Outcome: Number of Participants Who Discontinued Due to a TEAE
Description: An AE was any untoward medical occurrence in a clinical study participant. TEAEs were defined, within a dosing group, as AEs that started on or after the first dose of study treatment through 30 days after the last dose of study drug.
Time Frame: From first dose up to safety follow-up period (Week 28)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930
Number analyzed (Participants) | 2
Participants | 1

7. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Serious Adverse Event (TESAE)
Description: An AE was any untoward medical occurrence in a clinical study participant. TEAEs were defined, within a dosing group, as AEs that started on or after the first dose of study treatment through 30 days after the last dose of study drug.
  A serious adverse event (SAE) was an adverse event/reaction that results in any of the following outcomes:
  * Death
  * Is life-threatening (participant was at immediate risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe)
  * Requires participant hospitalization (formal admission to a hospital for medical reasons) or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity (ie, there was a substantial disruption of a person's ability to carry out normal life functions)
  * Is a congenital anomaly/birth defect
Time Frame: From first dose up to safety follow-up period (Week 28)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930
Number analyzed (Participants) | 2
Participants | 0

8. Secondary Outcome: Number of Participants Who Experienced a Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or 4 TEAE
Description: An AE was any untoward medical occurrence has no causal relationship with the study drug or with the clinical study itself. It was an unfavorable & unintended sign, symptom, syndrome, or illness that developed or worsened during clinical study.
  TEAEs: AEs that started on or after first dose of treatment through 30 days after the last dose of study drug. All AEs were graded using the CTCAE Grades 1 through 5.
  Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated
  Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL
  Grade 4: Life-threatening consequences; urgent intervention indicated
  Grade 5: Death
  Participants with Grades 3 or 4 AEs were reported
Time Frame: From first dose up to safety follow-up period (Week 28)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930
Number analyzed (Participants) | 2
Participants | 1

9. Secondary Outcome: Number of Participants Who Experienced a CTCAE Treatment-emergent Grade 3 or 4 Laboratory Abnormality
Description: Treatment-emergent Laboratory Abnormality were defined as an event that started on or after the first dose of study treatment through 30 days after the last dose of study drug.
  CTCAE Grades for laboratory abnormalities include:
  Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL.
  Grade 4: Life-threatening consequences; urgent intervention indicated.
  Grade 5: Death
  Participants with Grades 3 or 4 laboratory abnormality were reported.
Time Frame: From first dose up to safety follow-up period (Week 28)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: From first dose up to safety follow-up period (Week 28)
Description: Safety population
Arm/Group | BCX9930
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCX9930 (N=2)
Eyelid oedema (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (5)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
The sponsor decided to prematurely terminate the study due to changes in the competitive landscape. Due to low enrolment in the study (N=2) and early termination of both participants, very limited data were available for analyses. Therefore, only key efficacy endpoints (24-hour uPCR, 24-hour urine protein excretion, and eGFR) and safety were analyzed and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT05162066/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT05162066/SAP_001.pdf